CLINICAL TRIAL: NCT02038673
Title: An Open-label Phase I Study of Oral ASP5878 at Single and Multiple Doses in Patients With Solid Tumors
Brief Title: An Open-label Phase I Study of Orally Available Novel Small-molecule Fibroblast Growth Factor Receptors (FGFR) 1,2,3 and 4 Inhibitor, ASP5878 at Single and Multiple Doses in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5878-CL-0101
Record Dates: First submitted 2014-01-15; First posted 2014-01-16 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumors
Keywords: ASP5878; FGFR 1,2,3 and 4 inhibitor
MeSH Terms: interventions — ASP5878

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Dose escalation part 0.5 mg QD (Experimental): Oral
  Interventions: Drug: ASP5878
- Dose escalation part 1.0 mg QD (Experimental): Oral
  Interventions: Drug: ASP5878
- Dose escalation part 2.0 mg QD (Experimental): Oral
  Interventions: Drug: ASP5878
- Dose escalation part 2.0 mg BID (Experimental): Oral
  Interventions: Drug: ASP5878
- Dose escalation part 4.0 mg BID (Experimental): Oral
  Interventions: Drug: ASP5878
- Dose escalation part 6.0 mg BID (Experimental): Oral
  Interventions: Drug: ASP5878
- Dose escalation part 10.0 mg BID (Experimental): Oral
  Interventions: Drug: ASP5878
- Dose escalation part 20.0 mg BID (Experimental): Oral
  Interventions: Drug: ASP5878
- Dose escalation part 16.0 mg BID (Experimental): Oral
  Interventions: Drug: ASP5878
- Expansion part Urothelial Carcinoma (Experimental): Oral
  Interventions: Drug: ASP5878
- Expansion part Hepatocellular Carcinoma (Experimental): Oral
  Interventions: Drug: ASP5878
- Expansion part Squamous Cell Lung Carcinoma (Experimental): Oral
  Interventions: Drug: ASP5878

INTERVENTIONS:
Drug: ASP5878 — oral

SUMMARY:
The objectives of this study are to determine the tolerability, safety, pharmacokinetics (PK), pharmacodynamics (PD), and efficacy of oral ASP5878 in participants with solid tumors.

DETAILED DESCRIPTION:
This study consists of two parts. In the dose-escalation part, ASP5878 (orally available novel small-molecule FGFR 1,2,3 and 4 inhibitor, multiple dosing once-a-day (q.d.), multiple dosing twice-a-day (b.i.d.) or 5-day on/2-day off dosing twice-a-day (5on-2off)) is administered to participants with solid tumors in an increasing dose manner, and the tolerability, safety, pharmacokinetics (PK), pharmacodynamics (PD) and efficacy of ASP5878 are evaluated in these participants. Cycle 0 consists of 3 days and Cycle 1 and subsequent cycles consist of 28 days each in the dose-escalation part. In the expansion part, 16mg twice-a-day 5-day on/2-day off dose of ASP5878 (5on-2off) is administered to participants with solid tumors and safety, PK, PD and efficacy of ASP5878 are evaluated. The expansion part starts from Cycle 1 and each cycle consists of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor.
* Participant must meet at least one of the following criteria in the judgment of the investigator or sub-investigator:

  * Disease progression despite standard therapies
  * Progressive disease without any standard therapies established
  * Standard therapies are considered intolerable
* Eastern Cooperative Oncology Group performance status 0 or 1.
* Predicted life expectancy ≥ 12 weeks in the judgment of the investigator or sub-investigator.

Exclusion Criteria:

* Participant with ≥ Grade 2 (CTCAE v 4.0-JCOG) persistent symptoms and objective findings due to the toxicity attributable to prior treatment with antitumor effect (except alopecia).
* Participant who received a prior treatment intended for antitumor effect (medication, surgery, radiotherapy, etc.) within 4 weeks prior to the planned first day of study drug dosing (or participant who received mitomycin C or Nitrosourea within 6 weeks prior to the planned first day of study drug dosing).
* A major surgical procedure within 4 weeks prior to the planned first day of study drug dosing or a surgical procedure is planned during the course of the study.
* Participant who were treated with other investigational drug or medical device within 4 weeks prior to the planned first day of study drug dosing.
* Participant who has a history of organ transplantation.
* Participant with a brain metastasis with symptoms or requiring treatment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
Dose-escalation part and Expansion part: Safety assessed by Adverse Events (AEs) | Up to 18 months
  Until one of the discontinuation criteria is met.
Dose-escalation part and Expansion part:Safety assessed by Vital signs | Up to 18 months
  Blood pressure, pulse rate and body temperature, Until one of the discontinuation criteria is met.
Dose-escalation part and Expansion part:Safety assessed by Body weight | Up to 18 months
  Until one of the discontinuation criteria is met.
Dose-escalation part and Expansion part:Safety assessed by Laboratory tests | Up to 18 months
  Hematology, blood biochemistry, blood coagulation tests and urinalysis, until one of the discontinuation criteria is met.
Dose-escalation part and Expansion part:Safety assessed by 12-lead ECGs | Up to 18 months
  ECG: Electrocardiogram, until one of the discontinuation criteria is met.
Dose-escalation part and Expansion part: Ophthalmology | Up to 18 months
  Eyesight, funduscopy, slit lamp microscopy, and Optical Coherence Tomography, until one of the discontinuation criteria is met.
Dose-escalation part and Expansion part: Bone density measurement | Up to 18 months
  Until one of the discontinuation criteria is met.
Dose-escalation part and Expansion part: Computed tomography (CT) Imaging assessment | Up to 18 months
  Until one of the discontinuation criteria is met.
Expansion part only: Echocardiogram | Up to 18 months
  Until one of the discontinuation criteria is met.

SECONDARY OUTCOMES:
Dose-escalation part: Pharmacokinetics (PK) parameter of ASP5878 in plasma: Cmax | Day 1 at Cycle 0 and Day 5 (5on-2off) or 27 (q.d./b.i.d.) at Cycle 1
  Cmax: Maximum concentration, Cycle 0: single dose, Cycle 1: multiple dose after Cycle 0
Dose-escalation part:PK parameter of ASP5878 in plasma: tmax | Day 1 at Cycle 0 and Day 5 (5on-2off) or 27 (q.d./b.i.d.) at Cycle 1
  tmax: Time of Cmax
Dose-escalation part:PK parameter of ASP5878 in plasma: AUClast | Day 1 at Cycle 0 and Day 5 (5on-2off) or 27 (q.d./b.i.d.) at Cycle 1
  AUClast: Area under the concentration-time curve from the time of dosing extrapolated to the last measurable concentration
Dose-escalation part: PK parameter of ASP5878 in plasma: AUCinf | Day 1 at Cycle 0 and Day 5 (5on-2off) or 27 (q.d./b.i.d.) at Cycle 1
  AUCinf: Area under the concentration-time curve from the time of dosing extrapolated to time infinity
Dose-escalation part: PK parameter of ASP5878 in plasma: t1/2 | Day 1 at Cycle 0 and Day 5 (5on-2off) or 27 (q.d./b.i.d.) at Cycle 1
  t1/2: Terminal elimination half-life
Dose-escalation part: PK parameter of ASP5878 in plasma: CL/F | Day 1 at Cycle 0 and Day 5 (5on-2off) or 27 (q.d./b.i.d.) at Cycle 1
  CL/F: Apparent total systemic clearance
Dose-escalation part: PK parameter of ASP5878 in plasma: Vz/F | Day 1 at Cycle 0 and Day 5 (5on-2off) or 27 (q.d./b.i.d.) at Cycle 1
  Vz/F: Apparent volume of distribution during the terminal elimination phase
Dose-escalation part: PK parameter of ASP5878 in urine: Ae | Day 1 at Cycle 0 and Day 5 (5on-2off) or 27 (q.d./b.i.d.) at Cycle 1
  Ae: Amount of ASP5878 excreted into the urine
Dose-escalation part: PK parameter of ASP5878 in urine: CLR | Day 1 at Cycle 0 and Day 5 (5on-2off) or 27 (q.d./b.i.d.) at Cycle 1
  CLR: Renal clearance
Dose-escalation part: Pharmacodynamic (PD) parameter: Serum FGF23 concentrations | Day 1 at Cycle 0 and Day 5 (5on-2off) or 27 (q.d./b.i.d.) at Cycle 1
  FGF: Fibroblast Growth Factor
Dose-escalation part: PD parameter: Serum inorganic phosphorus concentrations | Day 1 at Cycle 0 and Day 5 (5on-2off) or 27 (q.d./b.i.d.) at Cycle 1
Dose-escalation part: PD parameter: Serum calcium concentrations | Day 1 at Cycle 0 and Day 5 (5on-2off) or 27 (q.d./b.i.d.) at Cycle 1
Dose-escalation part: PD parameter: Serum iPTH concentrations | Day 1 at Cycle 0 and Day 5 (5on-2off) or 27 (q.d./b.i.d.) at Cycle 1
  iPTH: Intact Parathyroid Hormone
Dose-escalation part: PD parameter: Serum calcitriol concentrations | Day 1 at Cycle 0 and Day 5 (5on-2off) or 27 (q.d./b.i.d.) at Cycle 1
Expansion part: PK parameter of ASP5878 in plasma: Cmax | Day 1 and 5 at Cycle 1
Expansion part: PK parameter of ASP5878 in plasma: tmax | Day 1 and 5 at Cycle 1
Expansion part: PK parameter of ASP5878 in plasma: AUClast | Day 1 and 5 at Cycle 1
Expansion part: PK parameter of ASP5878 in plasma: AUCinf | Day 1 and 5 at Cycle 1
Expansion part: PK parameter of ASP5878 in plasma: t1/2 | Day 1 and 5 at Cycle 1
Expansion part: PK parameter of ASP5878 in plasma: CL/F | Day 1 and 5 at Cycle 1
Expansion part: PK parameter of ASP5878 in plasma: Vz/F | Day 1 and 5 at Cycle 1
Expansion part: PD parameter: Serum FGF19 concentrations | Up to 18 months
  Until one of the discontinuation criteria is met.
Expansion part: PD parameter: Serum FGF23 concentrations | Up to 18 months
  Until one of the discontinuation criteria is met.
Expansion part: PD parameter: Serum inorganic phosphorus concentrations | Up to 18 months
  Until one of the discontinuation criteria is met.
Expansion part: PD parameter: Serum iPTH concentrations | Up to 18 months
  Until one of the discontinuation criteria is met.
Expansion part: PD parameter: Serum calcitriol concentrations | Up to 18 months
  Until one of the discontinuation criteria is met.
Expansion part: PD parameter: Serum 7α-hydroxy-4-cholesten-3-one | Up to 18 months
  Until one of the discontinuation criteria is met
Expansion part: Overall response | Up to 18 months
  Antitumor activity evaluated based on RECIST version 1.1, until one of the discontinuation criteria is met. Antitumor response is rated on a 4-level scale shown below (complete response [CR], partial response [PR], progressive disease [PD] and stable disease [SD]).
Expansion part: Maximum Shrinkage in Target Lesion | Up to 18 months
  Best percent change from baseline in the sum of diameters of all target lesions.
Expansion part: Progression free survival (PFS) | Up to 18 months
  Time from the start of the study treatment until death from any cause or Progressive Disease assessed according to RECIST 1.1.
Expansion part: Time to progression (TTP) | Up to 18 months
  Time from the start of the study treatment until Progressive Disease assessed according to RECIST 1.1.
Expansion part: Time to treatment failure (TTF) | Up to 18 months
  Time from the start of the study drug treatment until discontinuation of study drug treatment for any reason.
Expansion part: Overall survival (OS) | Up to 18 months
  Time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (35):
- United States (6):
  - Site US402, Orange, California
  - Site US401, New York, New York
  - Site US404, Cleveland, Ohio
  - Site US406, Spartanburg, South Carolina
  - Site US410, Fairfax, Virginia
  - Site US403, Seattle, Washington
- Japan (22):
  - Site JP122, Chiba
  - Site JP108, Fukuoka
  - Site JP115, Fukuoka
  - Site JP120, Fukuoka
  - Site JP116, Hokkaido
  - Site JP113, Hyōgo
  - Site JP103, Ibaraki
  - Site JP111, Ishikawa
  - Site JP119, Kanagawa
  - Site JP101, Kyoto
  - Site JP109, Miyagi
  - Site JP110, Miyagi
  - Site JP112, Nagoya
  - Site JP117, Niigata
  - Site JP121, Okayama
  - Site JP104, Osaka
  - Site JP106, Osaka
  - Site JP118, Osaka
  - Site JP124, Shizuoka
  - Site JP102, Tokyo
  - Site JP107, Tokyo
  - Site JP123, Tokyo
- South Korea (4):
  - Site KR202, Gyeonggi-do
  - Site KR201, Seoul
  - Site KR203, Seoul
  - Site KR204, Seoul
- Taiwan (3):
  - Site TW302, Tainan
  - Site TW301, Taipei
  - Site TW303, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=262